CLINICAL TRIAL: NCT06236893
Title: A Randomized, Double-Blind Placebo-Controlled Trial to Assess The Overall User Experience of a Synbiotic Vaginal Suppository
Brief Title: Randomized, Double-Blind Placebo-Controlled Trial to Assess Overall User Experience of a Synbiotic Vaginal Suppository
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seed Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20260
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Vaginal Personal Care
Keywords: Lactobacillus crispatus; vaginal malodor; vaginal discharge; vaginal itching; vaginal irritation; vaginal dryness
MeSH Terms: conditions — Vaginal Discharge

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VH-01 vaginal suppository tablet (Experimental): Participants will be instructed to take VH-01 vaginal suppository tablet (active product) as directed.
  Interventions: Other: VH-01 vaginal suppository tablet
- Placebo vaginal suppository tablet (Placebo Comparator): Participants will be instructed to take the placebo vaginal suppository tablet as directed. The placebo vaginal suppositories do not contain active ingredients and are identical in appearance to the active product.
  Interventions: Other: Placebo vaginal suppository tablet

INTERVENTIONS:
Other: VH-01 vaginal suppository tablet — Participants will be instructed to take VH-01 Days 1, 4, 7, 14, and 21 of Month 1 and Days 1 and 14 of Months 2 and 3.
  Arms: VH-01 vaginal suppository tablet
Other: Placebo vaginal suppository tablet — Participants will be instructed to take the placebo on Days 1, 4, 7, 14, and 21 of Month 1 and Days 1 and 14 of Months 2 and 3.
  Arms: Placebo vaginal suppository tablet

SUMMARY:
The purpose of this study is to assess the impact of a personal care product on vaginal health in individuals with a self-reported history of vaginal discomforts such as malodor, bothersome discharge, itching, irritation, and dryness. The personal care product, VH-01 contains a prebiotic and three distinct strains of Lactobacillus crispatus, a microbe commonly found in healthy vaginal microbiomes. The study will be a randomized, placebo-controlled trial where the test product will be compared to a placebo in a 2:1 manner. Participants will be asked to complete online questionnaires and provide vaginal samples to assess microbial communities.

The aims of this study are to assess:

1. The user experience and acceptability of VH-01 vaginal suppository vs. placebo.
2. Attitudes and perceptions of VH-01 vaginal suppository usage vs. placebo.
3. Health-related quality of life during the use of VH-01 vaginal suppository vs. placebo.
4. Changes in self-perceived vaginal discomforts during the use of VH-01 vaginal suppository vs. placebo.

DETAILED DESCRIPTION:
The vaginal microbiome is a community of microorganisms that live inside of the vagina. Studies have shown that vaginal microbiomes can be classified into one of five community state types (CSTs) known as: CST I, II, III, IV, and V. CSTs are determined based on the taxonomic composition of the vaginal microbiome. CST I, dominated by Lactobacillus crispatus, is considered optimal and is significantly associated with vaginal health.

Lactobacillus crispatus produces lactic acid and other compounds that maintain an optimal vaginal pH, which discourages the growth of harmful microbes that lead to disruptions in the vaginal microbial ecosystem. These disruptions may increase vaginal discomforts such as vaginal malodor, discharge, itching, irritation, and dryness.

VH-01 is a multi-strain vaginal synbiotic designed to seed and sustain an optimal and protective CST I vaginal ecology. The product delivers an ecology of complimentary Lactobacillus crispatus and synbiotic ingredients to promote an optimal vaginal ecology. The strains were selected to confer maximal vaginal microbiome stability in response to potential perturbations such as menstruation, sex, exercise, medication and other environmental influences.

The purpose of this study is to determine whether vaginal health can be influenced by a novel personal care product comprised of a prebiotic, and multiple strains of Lactobacillus crispatus associated with a stable vaginal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a vagina 18 - 55 years old at time of electronic consent
* Sex assigned female at birth
* Self-reported history of any of the following vaginal discomforts occurring recently and regularly, including but not limited to: Vaginal malodor, Bothersome vaginal discharge, Vaginal itching, Vaginal irritation, Vaginal dryness
* Willing to use an intra-vaginal suppository during the study and not knowing the product identity (active or placebo)
* Willing to complete questionnaires, which include questions related to vaginal health and sexual history/behavior
* Able to read and comprehend English and provide written informed consent
* Have reliable access to the internet

Exclusion Criteria:

* In menopause or experiencing menopausal symptoms
* History of irregular menses; defined as less than 25 day or more than 35 day cycle or length of time between cycles varies by more than 9 days
* Planned insertion or replacement of IUD in next 3 months (if applicable)
* Active pelvic or vaginal infection (i.e., active urinary tract infection, active bacterial vaginosis, active yeast infection). NOTE: Eligible to re-screen 4 weeks after completion of treatment for an active infection.
* Current or anticipated oral or vaginal antibiotic/antifungal treatment in the next 3 months (e.g., preoperative antibiotics for upcoming elective procedure). NOTE: Eligible to re-screen 4-weeks after completion of treatment
* Unwilling to discontinue the use of specified intra-vaginal products during the study including the following: vaginal probiotic suppositories, vaginal moisturizers, boric acid suppositories, pH balancing wipes, intravaginal gel, external vaginal itch relief cream, odor control sprays, vaginal steam products, vaginal cleansing douche, feminine/vaginal cleanser, vaginal preventive deodorant, gel/cream treatments for feminine odor
* Orally administered probiotics for vaginal health. NOTE: Oral probiotics for non-vaginal conditions (e.g., gastrointestinal health) are permitted. Eligible to re-screen 1-week after discontinuing orally administered probiotics for vaginal health
* Pregnant, breastfeeding or trying to conceive during the course of the study
* Active abnormal uterine/vaginal bleeding
* Receiving chronic oral steroid therapy (excluding those for skin, eyes, nose, or inhaled) or have received such therapy within 4 weeks of screening
* Surgery, immunotherapy, chemotherapy, radiation or biological cancer therapy within 30 days of enrollment and/or planned during the next 3 months
* Allergy to any components of the supporting or excipient ingredients in test formulation tablets/placebo
* Active serious medical condition requiring current treatment including but not limited to: Cancer, Autoimmune diseases (lupus, rheumatoid arthritis, Crohn's disease), Chronic infections (e.g., HIV, Hepatitis B, Hepatitis C), Serious cardiac, liver, or kidney disease, Psychiatric conditions/substance use disorders,
* Any condition which in the investigator's opinion may jeopardize the individual's safety or interfere with the ability to comply with the study
* Lives in the state of Alaska, Louisiana, New Jersey or New York

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
To evaluate user experience of VH-01 vaginal suppository vs. placebo. | From enrollment through three complete menstrual cycles or approximately 3 months.
  Self-reported rate of product acceptance to support vaginal health through month 3.

SECONDARY OUTCOMES:
To evaluate attitudes and perceptions of VH-01 vaginal suppository usage vs. placebo. | From enrollment through three complete menstrual cycles or approximately 3 months.
  Self-reported change in perception of vaginal state through month 3 [5-point Likert scale].
To evaluate health-related quality of life during the use of VH-01 vaginal suppository vs. placebo. | From enrollment through three complete menstrual cycles or approximately 3 months.
  Self-reported change in vaginal health-related quality of life through month 3 [5-point Likert scale].

OTHER OUTCOMES:
To evaluate changes in self-perceived vaginal discomforts during the use of VH-01 vaginal suppository vs. placebo. | From enrollment through three complete menstrual cycles or approximately 3 months.
  Self-reported change in specific vaginal discomforts through month 3 [10-point linear scale].

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Gevers, PhD, Study Director
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No